CLINICAL TRIAL: NCT00823758
Title: Understanding Patient's Knowledge and Use of Acetaminophen
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0577; 1U18HS017991-01 (AHRQ)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Liver Failure
Keywords: Acetaminophen; Liver; Centers for Education and Research on Therapeutics; CERTS; Over-the-counter Acetaminophen; OTC; Self-administration; Parental administration; Houston; Texas; Liver toxicity; Qualitative study; Pharmacists; Adolescents; Primary care physicians; Family Practitioners; General Internist
MeSH Terms: conditions — Liver Failure | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1: Parents of children under 8 years of age who have ever given their children an over- the-counter medication.
  Interventions: Behavioral: Focus Groups
- 2: Adolescents who are 13 to 20 years of age who have ever heard of over-the-counter medication.
  Interventions: Behavioral: Personal Interviews
- 3: Adults (21 years of age or older) who have used over-the-counter medication in the past 2 years.
  Interventions: Behavioral: Focus Groups
- 4: Primary care physicians will be Family Practitioners or General Internist, with an active Texas license, who devote at least 50% of their time to clinical practice.
  Interventions: Behavioral: Focus Groups
- 5: Pharmacists holding a PharmD degree and licensure in the state of Texas and work at least half-time in a community pharmacy setting.
  Interventions: Behavioral: Focus Groups

INTERVENTIONS:
Behavioral: Focus Groups — 6 to 8 participants per group.
  Groups: 1; 3; 4; 5
Behavioral: Personal Interviews — Conducted by phone and audiotaped.
  Groups: 2

SUMMARY:
Introduction to Study Objectives:

In a joint collaboration of the Centers for Education and Research on Therapeutics (CERTS) at The University of Pennsylvania and the M.D. Anderson Cancer Center, this study proposes to a) combine detailed but under-utilized existing large datasets and b) collect new primary data; together, resulting two data resources will advance our ability to describe, study, and understand the effectiveness and safety of pharmaceuticals received by pediatric patients in hospitals, and how to improve the safe use of over-the-counter (OTC) acetaminophen in home settings.

The CERTS study is organized into two projects: Project I and Project II.

For this protocol, the study focus will be Project II-Phase 1.

Project II will seek to qualitatively describe the patterns of use and misuse of over-the-counter OTC acetaminophen, through information gathered from consumers of various age groups, as well as professional key informants.

Project II-Phase 1

Objective 1:

-Qualitatively explore knowledge, attitudes, beliefs, and practices regarding adult and adolescent self-administration of OTC acetaminophen, and parental administration of OTC acetaminophen to children.

Objective 2:

-Qualitatively explore experiences and practices of key professional informants, including physician and pharmacists, with respect to communicating information on the administration and risks of OTC acetaminophen to consumers and patients.

DETAILED DESCRIPTION:
Individual Interviews:

If you agree to take part in this study, you will take part in individual interview session. The interviews will be conducted by phone and audiotaped (recorded) and transcribed (typed) by the research staff at M. D. Anderson.

You will be asked a series of questions about your knowledge of acetaminophen, views about the packaging, beliefs about the benefits and risks of taking acetaminophen, and when and how often you use acetaminophen. You will also be asked about what you have heard from other people about using acetaminophen and what types of experiences other people that you talked to about acetaminophen have had. The interview should last about 30 minutes.

To protect your confidentiality, only first names will be used during the interview sessions. Your name and any identifiable information will be removed when the audio recordings are typed. The audio recordings will be stored in a password protected file that only the study chair and research staff will have access to. The audio recordings will be destroyed by the researchers once study results have been published.

Length of Study:

Your participation in this study will be over after the interview is complete.

This is an investigational study.

Up to 124 people will be enrolled in this multicenter study. All will be enrolled by M. D. Anderson research staff. Participants will be recruited from outpatient pediatrics and primary care clinics at Kelsey-Seybold and Harris County Hospital District.

Focus Group Session:

The focus group session will be led by a trained interviewer. There will also be a research staff member present. During the focus group sessions, the interviewer will ask the group questions about acetaminophen, the directions on the packaging, beliefs about the benefits and risks of taking acetaminophen, and when and how often you use acetaminophen. Each focus group session should last about 90-120 minutes and will have 6-8 participants. The study chair will decide which focus group you will participate in.

You will take part in one of the following groups:

* Parents of children less than 8 years old will meet to talk about how acetaminophen is given to children.
* Adults will meet to talk about your beliefs about the benefits and risks of taking acetaminophen, how you take acetaminophen, and how often you take acetaminophen.

The focus group sessions will be audiotaped (recorded) and transcribed (typed) by the research staff at M. D. Anderson. To protect your confidentiality, only first names will be used during the focus group sessions and names will be coded when typed. The audio recordings will be destroyed by the researchers once study results have been published.

Length of Study:

Your participation on this study will be over when the focus group session is complete.

This is an investigational study. Up to 124 people will be enrolled in this multicenter study. All will be enrolled by M. D. Anderson research staff. Participants will be recruited from outpatient pediatrics and primary care clinics at Kelsey-Seybold and Harris County Hospital District.

ELIGIBILITY:
Inclusion Criteria:

1. English or Spanish language proficiency.
2. Residence in Metropolitan Houston, Texas.
3. Adequate cognition as determined by the research staff through the use of questions related to orientation about person, time and place.
4. Adolescents who are 13 to 20 years of age who have ever heard of over-the-counter medication (We will recruit 20 adolescents through their parents, who will be required to give consent before the study staff contacts the child);or parents of children (either a mother or a father, but only one parent per family) under 8 years of age who have ever given their children an over- the-counter medication; or adults (21 years of age or older) who have used over-the-counter medication in the past 2 years.
5. Primary care physicians will be Family Practitioners or General Internist, with an active Texas license, who devote at least 50% of their time to clinical practice.
6. Pharmacists will hold a PharmD degree and licensure in the state of Texas and work at least half-time in a community pharmacy setting.

Exclusion Criteria:

1. Participants who do not give informed consent.
2. A parent whose spouse/partner is/has already participated in the focus group.
3. Pharmacists actively enrolled in a training program.
4. Physicians who are participating in a fellowship or residency training program.
5. Children who may be depressed or at risk of suicide or managing that risk.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents of young children (8 years of age or younger) who administered acetaminophen to their children, Adults and Adolescents (aged 13-20 years of age) familiar with or used OTC acetaminophen in the last 2 years, and Primary care physicians and Pharmacists. All Houston, Texas residents.
Sampling Method: Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2008-12-19 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Qualitatively Described Patterns of Use + Misuse of Over-the-counter (OTC) Acetaminophen | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Maria Suarez-Almazor, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - The Children's Hospital of Philadelphia, University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Harris County Hospital District Outpatient Clinics, Houston, Texas
  - Kelsey Seybold, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org